CLINICAL TRIAL: NCT00004931
Title: A Clinical Trial Comparing 5-Fluorouracil (5-FU) Plus Leucovorin (LV) and Oxaliplatin With 5-FU Plus LV for the Treatment of Patients With Stages II and III Carcinoma of the Colon
Brief Title: Fluorouracil Plus Leucovorin With or Without Oxaliplatin in Treating Patients With Stage II or Stage III Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03165; NSABP-C-07; U10CA012027 (NIH)
Record Dates: First submitted 2000-03-07; First posted 2003-05-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Stage II Colon Cancer; Stage III Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Leucovorin; Fluorouracil; Oxaliplatin

ARMS (2):
- Arm I (Experimental): Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV (administered after 1 hour of leucovorin calcium) weekly for 6 weeks.
  Interventions: Drug: leucovorin calcium; Drug: fluorouracil; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 and leucovorin calcium and fluorouracil as in arm I.
  Interventions: Drug: leucovorin calcium; Drug: fluorouracil; Drug: oxaliplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
  Arms: Arm II
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Randomized phase III trial to compare the effectiveness of fluorouracil plus leucovorin with or without oxaliplatin in treating patients who have stage II or stage III colon cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective for colon cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the relative efficacy of 5-FU + LV + Oxaliplatin (FLOX) with that of 5-FU + LV (FL) in prolonging DFS.

SECONDARY OBJECTIVES:

I. To compare the relative efficacy of FLOX with FL in prolonging S.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

ARM I: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV (administered after 1 hour of leucovorin calcium) weekly for 6 weeks.

ARM II: Patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 and leucovorin calcium and fluorouracil as in arm I.

Treatment in both arms repeats every 8 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 6, 9, and 12 months; every 6 months for 4 years; and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must consent to be in the study and must have signed and dated an IRB-approved consent form conforming to federal and institutional guidelines
* In the opinion of the investigator, patients must have a 10-year life expectancy, excluding their diagnosis of cancer
* The interval between curative resection and randomization must be no more than 42 days
* The distal extent of the tumor must be >= 12 cm from the anal verge on endoscopy
* Patients must have colonic adenocarcinoma that meets one of the criteria below:

  * Stage II carcinoma (T3, 4; N0; M0) - The tumor invades through the muscularis propria into the subserosa, or into non-peritonealized pericolic or perirectal tissues (T3) or directly invades other organs or structures, and/or perforates visceral peritoneum (T4), excluding free perforation
  * Stage III carcinoma (any T; N1, 2; M0) - The tumor has invaded to any depth, with involvement of regional lymph nodes
* AGCs >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Bilirubin within or below the normal limits for the laboratory
* Alkaline phosphatase within or below the normal limits for the laboratory
* SGOT or SGPT within or below the normal limits for the laboratory
* Serum creatinine within or below the normal limits for the laboratory
* Patients with more than one synchronous primary colon tumor are eligible; for the purpose of this protocol, staging classification will be based on the stage of the more advanced primary tumor
* Patients are eligible if adjacent structures (e.g., bladder, small intestine, ovary, etc.) involved by direct extension of the primary tumor are removed en bloc and if, in the judgement of the surgeon and by confirmation on histological examination (i.e., margins of resection are not involved), the resection is deemed to be "curative"
* Patients must have an ECOG performance status of 0, 1, or 2
* Patients with intestinal obstruction are eligible; preliminary or complementary colostomy does not preclude entry
* Patients with prior noncolorectal malignancies are eligible if they have been disease-free for >= 5 years; patients with squamous or basal cell carcinoma of the skin that has been effectively treated, carcinoma in situ of the cervix that has been treated by operation only, or lobular carcinoma in situ of the breast are eligible, even if these conditions were diagnosed within 5 years prior to randomization

Exclusion Criteria:

* Prior invasive colon or rectal malignancy, regardless of disease-free interval
* Current or past malignant colon tumors other than carcinoma, i.e., sarcoma, lymphoma, carcinoid, etc., regardless of disease-free interval
* Tumors located < 12 cm from the anal verge on preoperative endoscopy
* Tumors that demonstrate free perforation as manifested by free air or free fluid in the abdomen; patients with walled-off perforation are eligible
* Pregnancy or lactation at the time of proposed randomization; (5-FU and oxaliplatin are both teratogenic and mutagenic and may cause fetal harm;) eligible patients of reproductive potential (both sexes) must agree to use adequate contraceptive methods
* Noncurative surgical resection or prior chemotherapy or radiotherapy for this malignancy, with the exception of a decompressing colostomy
* Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude the patient's receiving either chemotherapy treatment option; specifically excluded are patients with active ischemic heart disease (class III or class IV myocardial disease -- New York Heart Association) or a recent history of myocardial infarction (within 6 months), or current symptomatic arrhythmia

  * Class III: Patients with cardiac disease resulting in marked limitation of physical activity; such patients are comfortable at rest; less-than-ordinary physical activity causes fatigue, palpitation, dyspnea, or anginal pain
  * Class IV: Patients with cardiac disease resulting in inability to perform any physical activity without discomfort; symptoms of cardiac insufficiency or the anginal syndrome may be present even at rest
* Psychiatric or addictive disorders that would preclude obtaining informed consent
* Multiple primary tumors involving both the colon and the rectum that would preclude the patient's being classified as having only colon cancer
* Evidence of laparoscopically-assisted colectomy, unless patients are participating in the Intergroup Protocol INT 0146 or the Australasian, Multi-center, Prospective, Randomized, Clinical Study Comparing Laparoscopic and Conventional Open Surgical Treatments of Colon Cancer in Adults (ALCCaS)
* Isolated, distant, or noncontiguous intra-abdominal metastases, even if resected, will render the patient ineligible
* Clinically significant peripheral neuropathy at the time of randomization (defined in the NCI Common Toxicity Criteria [CTC] as grade 2 or greater neurosensory or neuromotor toxicity)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2472 (Estimated)
Dates: Start 2000-02; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
DFS rate | Time to first documented evidence of colon cancer recurrence, second primary cancer, or death from any cause without prior evidence of colon cancer recurrence or second primary cancer, assessed up to 3 years

SECONDARY OUTCOMES:
Survival rate | Time to death from any cause, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Kuebler, Principal Investigator — NSABP Foundation Inc
Locations (1):
- National Surgical Adjuvant Breast and Bowel Project, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Chen L, Wang Y, Cai C, Ding Y, Kim RS, Lipchik C, Gavin PG, Yothers G, Allegra CJ, Petrelli NJ, Suga JM, Hopkins JO, Saito NG, Evans T, Jujjavarapu S, Wolmark N, Lucas PC, Paik S, Sun M, Pogue-Geile KL, Lu X. Machine Learning Predicts Oxaliplatin Benefit in Early Colon Cancer. J Clin Oncol. 2024 May 1;42(13):1520-1530. doi: 10.1200/JCO.23.01080. Epub 2024 Feb 5. PMID 38315963
- [Derived] Cohen R, Taieb J, Fiskum J, Yothers G, Goldberg R, Yoshino T, Alberts S, Allegra C, de Gramont A, Seitz JF, O'Connell M, Haller D, Wolmark N, Erlichman C, Zaniboni A, Lonardi S, Kerr R, Grothey A, Sinicrope FA, Andre T, Shi Q. Microsatellite Instability in Patients With Stage III Colon Cancer Receiving Fluoropyrimidine With or Without Oxaliplatin: An ACCENT Pooled Analysis of 12 Adjuvant Trials. J Clin Oncol. 2021 Feb 20;39(6):642-651. doi: 10.1200/JCO.20.01600. Epub 2020 Dec 23. PMID 33356421
- [Derived] Salem ME, Yin J, Goldberg RM, Pederson LD, Wolmark N, Alberts SR, Taieb J, Marshall JL, Lonardi S, Yoshino T, Kerr RS, Yothers G, Grothey A, Andre T, De Gramont A, Shi Q. Evaluation of the change of outcomes over a 10-year period in patients with stage III colon cancer: pooled analysis of 6501 patients treated with fluorouracil, leucovorin, and oxaliplatin in the ACCENT database. Ann Oncol. 2020 Apr;31(4):480-486. doi: 10.1016/j.annonc.2019.12.007. Epub 2020 Jan 16. PMID 32085892
- [Derived] Taieb J, Shi Q, Pederson L, Alberts S, Wolmark N, Van Cutsem E, de Gramont A, Kerr R, Grothey A, Lonardi S, Yoshino T, Yothers G, Sinicrope FA, Zaanan A, Andre T. Prognosis of microsatellite instability and/or mismatch repair deficiency stage III colon cancer patients after disease recurrence following adjuvant treatment: results of an ACCENT pooled analysis of seven studies. Ann Oncol. 2019 Sep 1;30(9):1466-1471. doi: 10.1093/annonc/mdz208. PMID 31268130
- [Derived] Song N, Pogue-Geile KL, Gavin PG, Yothers G, Kim SR, Johnson NL, Lipchik C, Allegra CJ, Petrelli NJ, O'Connell MJ, Wolmark N, Paik S. Clinical Outcome From Oxaliplatin Treatment in Stage II/III Colon Cancer According to Intrinsic Subtypes: Secondary Analysis of NSABP C-07/NRG Oncology Randomized Clinical Trial. JAMA Oncol. 2016 Sep 1;2(9):1162-9. doi: 10.1001/jamaoncol.2016.2314. PMID 27270348
- [Derived] Yothers G, O'Connell MJ, Lee M, Lopatin M, Clark-Langone KM, Millward C, Paik S, Sharif S, Shak S, Wolmark N. Validation of the 12-gene colon cancer recurrence score in NSABP C-07 as a predictor of recurrence in patients with stage II and III colon cancer treated with fluorouracil and leucovorin (FU/LV) and FU/LV plus oxaliplatin. J Clin Oncol. 2013 Dec 20;31(36):4512-9. doi: 10.1200/JCO.2012.47.3116. Epub 2013 Nov 12. PMID 24220557
- [Derived] Yothers G, Sargent DJ, Wolmark N, Goldberg RM, O'Connell MJ, Benedetti JK, Saltz LB, Dignam JJ, Blackstock AW; ACCENT Collaborative Group. Outcomes among black patients with stage II and III colon cancer receiving chemotherapy: an analysis of ACCENT adjuvant trials. J Natl Cancer Inst. 2011 Oct 19;103(20):1498-506. doi: 10.1093/jnci/djr310. Epub 2011 Oct 12. PMID 21997132
- [Derived] Yothers G, O'Connell MJ, Allegra CJ, Kuebler JP, Colangelo LH, Petrelli NJ, Wolmark N. Oxaliplatin as adjuvant therapy for colon cancer: updated results of NSABP C-07 trial, including survival and subset analyses. J Clin Oncol. 2011 Oct 1;29(28):3768-74. doi: 10.1200/JCO.2011.36.4539. Epub 2011 Aug 22. PMID 21859995
- [Derived] Fumagalli D, Gavin PG, Taniyama Y, Kim SI, Choi HJ, Paik S, Pogue-Geile KL. A rapid, sensitive, reproducible and cost-effective method for mutation profiling of colon cancer and metastatic lymph nodes. BMC Cancer. 2010 Mar 16;10:101. doi: 10.1186/1471-2407-10-101. PMID 20233444
- [Derived] Kuebler JP, Colangelo L, O'Connell MJ, Smith RE, Yothers G, Begovic M, Robinson B, Seay TE, Wolmark N. Severe enteropathy among patients with stage II/III colon cancer treated on a randomized trial of bolus 5-fluorouracil/leucovorin plus or minus oxaliplatin: a prospective analysis. Cancer. 2007 Nov 1;110(9):1945-50. doi: 10.1002/cncr.23013. PMID 17853393
- [Derived] Kuebler JP, Wieand HS, O'Connell MJ, Smith RE, Colangelo LH, Yothers G, Petrelli NJ, Findlay MP, Seay TE, Atkins JN, Zapas JL, Goodwin JW, Fehrenbacher L, Ramanathan RK, Conley BA, Flynn PJ, Soori G, Colman LK, Levine EA, Lanier KS, Wolmark N. Oxaliplatin combined with weekly bolus fluorouracil and leucovorin as surgical adjuvant chemotherapy for stage II and III colon cancer: results from NSABP C-07. J Clin Oncol. 2007 Jun 1;25(16):2198-204. doi: 10.1200/JCO.2006.08.2974. Epub 2007 Apr 30. PMID 17470851